CLINICAL TRIAL: NCT03489616
Title: Chemotherapy Combination With Local Radiotherapy and rhGM-CSF for Oligometastatic Stage IV NSCLC Patients Without Progression After First-line Chemotherapy: a Prospective Randomized Controlled Study
Brief Title: Chemotherapy Combination With Local Radiotherapy and rhGM-CSF for Oligometastatic Stage IV NSCLC Patients
Acronym: CRAGMOLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, chief physician, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDCH201701LC
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — regramostim; sargramostim; Pemetrexed; Pharmaceutical Preparations; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy+chemotherapy+ rhGM-CSF (Experimental): Patients with PR or SD after first-line chemotherapy will be treated with pemetrexed on d1 (500mg/m2) or other single agent on d1, d8. Local radiotherapy dose will be> 4Gy per time（or BED >45Gy） from day 2 to day 15 in a cycle of 21 days. Subcutaneous injection of rhGM-CSF (200ug/m² per day) will be executed 24 hours after chemotherapy. Repeat in the second metastatic lesions.
  Interventions: Biological: rhGM-CSF; Drug: Pemetrexed; Radiation: Local Radiotherapy; Drug: Single agent
- Single agent maintenance therapy (Experimental): Maintenance treatment by single agent in a cycle of 21 days.
  Interventions: Drug: Single agent

INTERVENTIONS:
Biological: rhGM-CSF — rhGM-CSF is a stimulator of the growth and differentiation of hematopoietic progenitor cells committed to neutrophils, monocytes or eosinophils. rhGM-CSF can promote the maturation of dendritic cells and macrophage, increase their antigen presentation ability.
  Other Names: Recombinant human granulocyte macrophage stimulating factor
  Arms: Radiotherapy+chemotherapy+ rhGM-CSF
Drug: Pemetrexed — Pemetrexed (brand name Alimta) is a chemotherapy drug manufactured and marketed by Eli Lilly and Company. Its indications are the treatment of pleural mesothelioma and non-small cell lung cancer.
  Arms: Radiotherapy+chemotherapy+ rhGM-CSF
Radiation: Local Radiotherapy — Radiotherapy promotes the release of tumor antigen
  Other Names: Local Radiation therapy
  Arms: Radiotherapy+chemotherapy+ rhGM-CSF
Drug: Single agent — Other chemotherapy drugs,such as Docetaxel, gemcitabine
  Other Names: Single agent for maintenance therapy

SUMMARY:
The purpose of this study is to determine whether chemotherapy combination with local radiotherapy and rhGM-CSF is safe, effective in the treatment of oligometastatic stage IV NSCLC patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether chemotherapy combination with local radiotherapy and recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) is safe, effective in the treatment of oligometastatic stage IV NSCLC patients who were PR or SD after first-line chemotherapy，and to observe the abscopal effect, whether the scheme can improve PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV NSCLC patients without clear driving genes who were PR or SD after standard first-line chemotherapy;
2. Patients who were oligometastasis evaluated by PET-CT or other examinations after first-line chemotherapy. Eligible patients should have 2 to 5 distant metastases (at least 2 metastases were suitable for low fractionated radiotherapy). At least one distant measurable lesion outside the radiation sites.
3. Age varied from 18 to 75 years old.
4. ECOG performance status 0-2.
5. Expected lifespan ≥3 months.
6. Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin ≥90 g/L.
7. Able to understand and give written informed consent and comply with study procedures.

Exclusion criteria

1. Allergy of rhGM-CSF and its accessories.
2. Disease of systemic immune or immune disorders.
3. Histology confirmed small cell carcinoma or other malignant compositions in the cancer tissue.
4. Patients with thrombotic disease or platelets ≥600×109/L
5. Cancer history within 5 years apart from NSCLC before enrollment.
6. Tumor related immunotherapy within 4 weeks, including but not limited to immune cell therapy, tumor vaccine therapy, Immune checkpoint therapy, and other immunomodulators (such as thymosin, lentinan) except for rhGM-CSF.
7. The abnormality of kidney , heart or lung functions（serum creatinine, Cr>177mol/L; serum AST or ALT more than 2 times above normal limits; total bilirubin, TBIL>34mol/L）.
8. HIV virus, hepatitis C virus or T lymphocyte virus (type1 or type 2) infection and active hepatitis or other uncontrolled infections.
9. Women in pregnancy or lactation.
10. Others who do not meet the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-Free-Survival

SECONDARY OUTCOMES:
Abscopal effect rate | At the time point of 4 weeks after completion of rhGM-CSF
  Radiotherapy-induced immune-mediated tumour regression at sites distant to the irradiated field
OS | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: JINMING YU, doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (2):
- China (2):
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - SHANDONG Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Result] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196